CLINICAL TRIAL: NCT04567381
Title: An Evaluation of the Project CHANGE-MS Violence Intervention Program
Brief Title: An Outcome Evaluation of the Project CHANGE-MS Violence Intervention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-165
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Violence; Recidivism
Keywords: Violence prevention; Hospital based; Community Violence; Violent Recidivism
MeSH Terms: conditions — Recidivism | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized into two separate groups, treatment as usual and enhanced services. Groups will be followed concurrently for one year for the outcomes of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (Active Comparator): Treatment as Usual (TAU)/Control. Individuals randomized to TAU will receive a list of resources which provides participants with community agency information that they can engage on their own. The list of resources will include contact information for various services such as housing, employment, mental health and legal services. Patients randomized into this condition receive little to no assistance from program staff and must navigate the vast terrain of social service providers on their own.
  Interventions: Other: Treatment as Usual
- Enhanced Services (Experimental): Enhanced Services/Treatment (ES). Participants randomized to the ES intervention will receive intensive community-based case management.
  Interventions: Other: Enhanced Services

INTERVENTIONS:
Other: Enhanced Services — In enhanced services, the provision of services go beyond just referring a patient and leaving them to follow-through on their own accord. ES varies based on resources, model of service delivery, philosophy, and role and responsibilities of team members. Enhanced services usually includes longer-term case management which can then facilitate the connection to clinical counseling, victim assistance, familial assistance, legal assistance, emergency financial funding, transportation for subsequent appointments related to a patient's medical condition, employment assistance, and assistance in educational program enrollment.
  Arms: Enhanced Services
Other: Treatment as Usual — Individuals randomized to TAU will receive a list of resources which provides participants with community agency information that they can engage on their own. The list of resources will include contact information for various services such as housing, employment, mental health and legal services. Patients randomized into this condition receive little to no assistance from program staff and must navigate the vast terrain of social service providers on their own.
  Arms: Treatment as Usual

SUMMARY:
This is a prospective randomized control trial design to evaluate the effectiveness of a hospital based violence intervention program. Participants will be randomized into a "treatment as usual" group who will receive written referrals for services and an "enhanced services" group who will receive intensive case management over a one year period. Primary outcome will be rate of violent reinjury after enrollment. Follow-up will be for one year.

DETAILED DESCRIPTION:
Potential study participants are all adult, male survivors of community violence treated at the study site.

After a potential study participant is screened and deemed eligible for participation in the study consent will be obtained to participate in the study. At stage one a participant can either accept or refuse services and at stage two can consent or refuse to consent in the study.

If a patient consents to both receive services and participate in the study, the participant will be randomly assigned to either the "Treatment as Usual" (TAU) intervention, which receives the referral card for services, or the "Enhanced Treatment" (ET) intervention prior to assessment so that the results of the assessment do not influence program staff which group the potential study participant is assigned. At the beginning of the study, 400 identical envelopes will be created, 200 with a slip of paper labeled "Treatment as Usual" and 200 with a slip of paper labeled "Enhanced Treatment." These will be shuffled and will be used to assign the random group of those patients that consent to participate.

Those who refuse services and refuse the study will not be included in the study. Finally, those who accept services but refuse to be in the study will not be in the study.

Participation in the study will take place in five stages. At stage one, after consenting to the study and being randomly assigned to TAU or ET care groups, the patient will undergo an interview. The interview will take place at bedside granted that privacy can be guaranteed or in an office if the patient is mobile. In some cases it may be appropriate to set up an appointment after discharge to conduct the interview. Patients that agree to participate in the study will be entered into a secure Excel Database on a MedStar password protected server. Only study personnel will have access to this database, which will contain a key with patient name and a unique identifier. This database will also be used to assess study quality measures of approaches to eligible participants and percent uptake. This database and the signed consents will have identifiable patient information. An additional SpreadSheet Web tool, provided by the DC Department of Health Office of Victims Services and Justice Grants will be used to track outcomes and follow-up of participants. This will include only de-identified information. The internal secure Excel database will have a link between patient name and unique identifier.

At stage two, the participant engages the project depending on which group they are in. Those in the ET group will receive a case manager whereas those in the TAU group will receive a referral card. Those in the ET will receive case management services and receive information and other counseling services whereas those who receive the referral card will be expected to engage the services on the referral cards provided.

At stage three, the study participants will be asked to conduct a smaller interview at month 6 after entry into the program to determine subsequent injury. The results of this interview will be recorded in the DC DOH-OVSJG SpreadSheet Web tool. In addition, partnership with CRISP (Chesapeake Regional Information System for our Patients) will be used to actively query whether or not participants have been seen in regional hospitals, EDs, or outpatient settings for repeat violent injury.

CRISP is a regional health information system and is entirely HIPAA compliant and has health information level security. It has been designated as Maryland's statewide health information exchange. Under a contract with CRISP, each site will be able to securely submit the names of patients that have agreed to participate in research. CRISP will then send notifications of patient care and each site will be able to have accurate follow-up of the main outcome (recidivism). This will allow validation of answers from telephone interviews at 6 and 12 months as well as gain accurate information on those participants that may be lost to follow-up. Patient information is relayed securely using specially designed HIPAA and confidentiality compliant email addresses, created for this purpose. All participants will specifically be asked for their permission to access CRISP for this purpose.

At stage four, approximately twelve months after entry into the study, the study participants will be engaged in the post-interview. Answers to this post-interview will be recorded and tracked in the DC DOH OVSJG SpreadSheet Web de-identified database.

Stage five will entail an invitation to a focus group. Four focus groups will be conducted after the quantitative data collection. Two of the focus groups will focus on those who have not successfully completed the program and two more will randomly sample among those who have successfully completed the program. The four focus groups will have no more than seven individuals. Focus groups will be conducted in a private, unlabeled conference room at the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. identify as male
2. be 18 years of age or older
3. speak English
4. have experienced a violent injury in the form of a gunshot wound, stabbing, or assault within two years of first contact with the program (verified through trauma registry)
5. experienced the injury within the borders of the east coast city where the study is taking place.

Exclusion Criteria:

1. identifying as female
2. reporting an age ≤ 17
3. experiencing a self-inflicted violent injury
4. experiencing a traumatic brain injury
5. being under police custody
6. not being injured within the borders of the east coast city where the study is taking place
7. not being able to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identified men
Enrollment: 400 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of violent reinjuries in 12 months | 12 months
  Subsequent violent reinjury
Number of participants with death in 12 months | 12 months
  Death

SECONDARY OUTCOMES:
Decreased in Frequency of Substance Abuse in past-30 days | 12 months
  Substance Abuse in previous 30 days from survey
Improvement of Level of Mastery as measured using Pearlin Mastery Scale | 12 months
  Extent one regards one's life-chances as being under one's own control
Improvement in Disposition towards Violence as measured using the Code of the Street Scale | 12 months
  Extent to which it is justifiable or advantageous to use violence using Simon's Code of the Street
Decrease in number of Medical Legal Needs screened positive | 12 months
  Number of screening civil medical legal needs
Improved Life Satisfaction | 12 months
  Measured with the Satisfaction with Life Scale, a 7-point Likert scale questionnaire with minimum score of 5, maximum of 35
Decreased Post-Traumatic Stress Disorder (PTSD) Symptoms measured using PTSD-8: A Short PTSD Inventory | 12 months
  measured using PTSD-8, an 8 question with 4-point Likert scale validated screening questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No